CLINICAL TRIAL: NCT03228277
Title: Phase II, Multicenter, Single-arm, Open-label Study to Evaluate the Efficacy of Olmutinib(Olita®) in Patients With NSCLC Who Harboring T790M Mutation Confirmed Using DNA Extracted From Extracellular Vesicles in Bronchoalveolar Lavage Fluid
Brief Title: Olmutinib Trial in T790M (+) NSCLC Patients Detected by Liquid Biopsy Using BALF Extracellular Vesicular DNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Kye Young Lee, Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KASTT005_BAL_Olita
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Extracellular vesicles; Bronchoalveolar lavage fluid; Liquid biopsy; T790M; NSCLC; Exosomes; EGFR mutation testing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — olmutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olmutinib (Experimental): Single arm of Olmutinib, staring dose of 800 mg
  Interventions: Drug: Olmutinib

INTERVENTIONS:
Drug: Olmutinib — Patients to be provided with Olmutinib 800mg (2 x 400 mg tablets) once daily (QD)
  Other Names: Olita®

SUMMARY:
The purpose of this study is to evaluate the efficacy of Olmutinib(Olita®) in patients with T790M-positive non-small cell lung cancer (NSCLC) confirmed using DNA extracted from extracellular vesicles of bronchoalveolar lavage fluid.

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase 2 study to assess the anti-tumor efficacy of Olmutinib(Olita®) administered to patients with T790M-positive NSCLC confirmed using DNA extracted from extracellular vesicles in bronchoalveolar lavage fluid as measured by objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 19 years
2. Obtained written informed consent
3. Histologically- or cytologically confirmed diagnosis of unresectable Stage IIIB or IV non-small cell lung cancer.
4. Confirmation that the tumor harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
5. Eastern Cooperative Oncology Group performance status of 0 to 2
6. Prior treatment with at least one line of a single agent EGFR TKI (gefitinib, erlotinib, afatinib) and confirmed progressive disease after treatment with EGFR TKI

   * Regardless of treatment sequence between previous chemotherapy and EGFR TKI
   * Regardless of whether they were administered conventional chemotherapy, if therapy were treated with at least one EGFR TKI
7. Subjects who will undergo bronchoscopy/ BAL procedures and sufficient amount of BAL fluid is carefully collected for EGFR mutation analysis.
8. Confirmation that the extracellular vesicles (EV) extracted from bronchoalveolar lavage fluid (BALF) harbour T790M mutation (It can be replaced previous the same result throughout the follow up period before enrollment.)
9. At least one measurable disease (except brain) at baseline according to RECIST version 1.1
10. Female subjects must be postmenopausal (for at least one year), or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and, for those of childbearing potential, have a negative urinary β-hCG pregnancy test at screening.
11. Male subjects should be willing to use barrier methods which are suitable for sexual partner throughout the study.
12. Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. The subject also must sign and date the consent form before specific procedures or sampling.
13. Adequate organ function as defined by liver, kidney, and hematologic laboratory testing as below

    * Absolute neutrophil count (ANC) ≥ 1500/mm3, Platelet ≥ 100,000 /mm3 Hemoglobin (Hb) ≥ 9.0g/dL
    * Serum creatinine ≤ upper limit of normal (ULN)
    * AST/ALT/ALP ≤ 3 times ULN, Total bilirubin ≤2.0 mg/dL AST/ALT/ALP ≤ 5 times ULN in patients with metastatic lesions to the liver ALP ≤ 5 times ULN in patients with metastatic lesions to the bone
14. Expected survival of at least 12 weeks

Exclusion Criteria:

1. Previous treatment with anticancer therapies, EGFR-TKI, olmutinib (HM61713), or other drugs that target T790M-positive mutant EGFR with sparing of wild-type, Osimertinib (AZD9291), Rociletinib (CO-1686), investigational agent(s) within 30 days prior to the first administration of study drug, radiotherapy
2. Treatment with a potent cytochrome P450 (CYP) 3A4 inhibitors or inducers
3. History of any other malignancy EXCEPTIONS are:

   * adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, thyroid cancer
   * other malignancies diagnosed prior to randomisation and treated with no evidence of disease recurrence more than 3 years
4. Any history or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of III or IV, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to enrolment. Increased QTc interval > 450 ms on screening ECG
5. Any history of presence of interstitial lung disease
6. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption).
7. Ongoing active infection with, hepatitis B virus (infection defined as a positive HbsAg and/ or HBV DNA), hepatitis C virus (infection defined as a positive HCV RNA), or human immunodeficiency virus (HIV) Type 1/2 infection at the time of screening.
8. Known history of hypersensitivity to active or inactive excipients of study drug (olmutinib) or drugs with a similar chemical structure of olmutinib
9. Subjects with galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
10. Symptomatic or uncontrolled central nervous system (CNS) metastases (Patients are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically and radiologically stable)
11. Uncontrolled active infectious disease (with the exception of those that are considered to be needed topical antibiotics, however subjects can be enrolled into the study after they complete their treatment)
12. Unable to attend all the study visits or comply with study procedures
13. Patients who had received other investigational product within 30 days prior to the first administration of study drug except for gefitinib, erlotinib, or afatinib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Change from baseline at every 6 weeks until disease progression or withdrawal from study, assessed up to 12 months
  defined as the proportion of patients who achieved complete remission(CR) or partial remission(PR) based on RECIST version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Change from baseline at every 6 weeks until disease progression or withdrawal from study, assessed up to 12 months
  defined as the proportion of patients with a documented CR, PR, and SD during the treatment cycles according to the RECIST version 1.1
Progression-free survival (PFS) | Change from baseline at every 6 weeks until disease progression or withdrawal from study, assessed up to 12 months
  defined as the time from first administration of study drug to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Kye Young Lee, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No